CLINICAL TRIAL: NCT04113317
Title: The Role of Granulocyte-Colony Stimulating Factor (G-CSF) for Improving PELD Score and Nutritional Status in Pediatric Liver Cirrhosis Prior to Liver Transplantation Through Immunomodulation of Neutrophil, CD34+ Cell, TNF-α and IL-10
Brief Title: Granulocyte-Colony Stimulating Factor (G-CSF) as Optimizing Therapy for Pediatric Liver Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Collaborators: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Tri Hening Rahayatri, Principal Investigator, Fakultas Kedokteran Universitas Indonesia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FakultasKUI
Record Dates: First submitted 2019-09-22; First posted 2019-10-02 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Liver Cirrhosis; Severe Malnutrition; PELD; Undernutrition
MeSH Terms: conditions — Liver Cirrhosis; Malnutrition | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Group (Experimental): Subcutaneous injection of G-CSF with dose of 5μg/kg/day for 5 days consecutively, in addition to a single dose every 3 days up to 12 times, as well as liver cirrhosis standard regimen
  Interventions: Drug: G-CSF (Filgrastim)
- Control Group (No Intervention): Liver cirrhosis standard treatment only

INTERVENTIONS:
Drug: G-CSF (Filgrastim) — Contains 0,59 mg of acetate, 0,04 mg of polysorbate 80, 0,035 mg of sodium, 50 mg of sorbitol
  Other Names: Neupogen
  Arms: Treatment Group

SUMMARY:
This study compares the effect of human recombinant Granulocyte-Colony Stimulating Factor (G-CSF) in pediatric patients with liver cirrhosis with a control group. The study aims to observe improvement of (Pediatric End-stage Liver Disease) PELD score and nutritional status prior to liver transplantation procedure. In addition to the intervention, standard treatments for liver cirrhosis are also given for both groups. G-CSF is administered for 12 times.

Condition of disease:

Pediatric patient aged 3 months to 12 years old Liver cirrhosis Undernourished / Severe malnutrition PELD score 10-25

Intervention:

Drug: Recombinant Human G-CSF

Phase:

Phase 3

DETAILED DESCRIPTION:
This open-label randomized control trial conducted in Cipto Mangunkusumo Hospital, Jakarta, Indonesia, aimed to determine the effect of G-CSF to improve PELD score and nutritional status of pediatric patients with liver cirrhosis prior to liver transplantation. A total of 52 pediatric patients with liver cirrhosis, malnutrition and PELD score between 10-25 will be collected and divided into intervention group and control group. The intervention group will be given a subcutaneous injection of G-CSF 5μg/kg/day for 5 days consecutively, followed by a single dose every 3 days up to 12 times throughout the trial. Additionally, both the intervention and control group receive standard liver cirrhosis treatment. Randomization is done using block randomization.

The patients will be clinically monitored and evaluated for anthropometric changes (body weight, mid-arm circumference, mid-arm muscle circumference, and triceps skinfold thickness), complete blood count, absolute neutrophil count, liver function tests, cytokines (IL-10, TNF-α), Procalcitonin, hepatocyte growth factor (HGF), CD34+ cell count and PELD score (albumin, bilirubin, prothrombin and international normalized ratio values).

Data analysis will be performed using IBM SPSS Statistics version 20.0.0.

ELIGIBILITY:
Inclusion Criteria:

* Age between 3 months to 12 years old
* Conscious state
* Without the presence of fever (temperature: <37,5°C)
* Decompensated liver cirrhosis
* Liver cirrhosis due to various etiology
* Undernourished or severe malnutrition
* PELD score between 10-25

Exclusion Criteria:

* Malignancy (liver origin or other types)
* History of undergoing any organ transplantation procedure
* Acute liver failure
* Failure of any organ other than the liver
* Encephalopathy
* Severe infection such as bacterial peritonitis and pneumonia

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
PELD Score | 90 days
  The scoring determines the individual's need for liver transplant. Calculation is based on an equation that incorporates the values of bilirubin serum, international normalized ratio, albumin and body growth measurement. Score ranges between 6 (low illness level) to 40 (severely ill).
Anthropometric Changes | 90 days
  Measurement of mid-arm circumference (MAC) will be obtained in centimeters and be plotted on the curve to observe changes in nutritional status

SECONDARY OUTCOMES:
Pro-inflammatory Marker | 30 days
  Tumor necrosis factor alpha (TNF-α) cytokine level in the blood will be the parameter for pro-inflammatory marker
Anti-inflammatory Marker | 30 days
  Interleukin-10 (IL-10) cytokine level in the blood will be the parameter for anti-inflammatory marker
Liver Regeneration Marker | 30 days
  hepatocyte growth factor (HGF) serum level will be the biochemical parameter for liver regeneration

CONTACTS AND LOCATIONS:
Overall Officials: Tri Hening Rahayatri, MD, Study Chair — Faculty of Medicine, Universitas Indonesia - Cipto Mangunkusumo Hospital; Akmal Taher, Study Director — Faculty of Medicine, Universitas Indonesia - Cipto Mangunkusumo Hospital
Locations (1):
- Fakultas Kedokteran Universitas Indonesia, Jakarta, Java, Indonesia

REFERENCES:
- [Background] Fioredda F, Lanza T, Gallicola F, Riccardi F, Lanciotti M, Mastrodicasa E, Signa S, Zanardi S, Calvillo M, Dufour C. Long-term use of pegfilgrastim in children with severe congenital neutropenia: clinical and pharmacokinetic data. Blood. 2016 Oct 27;128(17):2178-2181. doi: 10.1182/blood-2016-07-727891. Epub 2016 Sep 12. No abstract available. PMID 27621310
- [Background] Dale DC, Crawford J, Klippel Z, Reiner M, Osslund T, Fan E, Morrow PK, Allcott K, Lyman GH. A systematic literature review of the efficacy, effectiveness, and safety of filgrastim. Support Care Cancer. 2018 Jan;26(1):7-20. doi: 10.1007/s00520-017-3854-x. Epub 2017 Sep 22. PMID 28939926
- [Background] Yang Q, Yang Y, Shi Y, Lv F, He J, Chen Z. Effects of Granulocyte Colony-Stimulating Factor on Patients with Liver Failure: a Meta-Analysis. J Clin Transl Hepatol. 2016 Jun 28;4(2):90-6. doi: 10.14218/JCTH.2016.00012. Epub 2016 Jun 15. PMID 27350939
- [Background] Garg V, Garg H, Khan A, Trehanpati N, Kumar A, Sharma BC, Sakhuja P, Sarin SK. Granulocyte colony-stimulating factor mobilizes CD34(+) cells and improves survival of patients with acute-on-chronic liver failure. Gastroenterology. 2012 Mar;142(3):505-512.e1. doi: 10.1053/j.gastro.2011.11.027. Epub 2011 Nov 23. PMID 22119930
- [Background] Chavez-Tapia NC, Mendiola-Pastrana I, Ornelas-Arroyo VJ, Norena-Herrera C, Vidana-Perez D, Delgado-Sanchez G, Uribe M, Barrientos-Gutierrez T. Granulocyte-colony stimulating factor for acute-on-chronic liver failure: systematic review and meta-analysis. Ann Hepatol. 2015 Sep-Oct;14(5):631-41. PMID 26256891